CLINICAL TRIAL: NCT00095095
Title: Lumbar Interbody Fusion Using The Telamon® Peek™ Versus The Telamon® Hydrosorb™ Fusion Device - A Prospective, Randomized Controlled Trial To Assess Surgical And Clinical Outcomes
Brief Title: Lumbar Interbody Fusion Using the Telamon® Peek™ Versus the Telamon® Hydrosorb™ Fusion Device
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Medtronic Spinal and Biologics (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL04-90
Record Dates: First submitted 2004-10-29; First posted 2004-11-01 (Estimated); Last update posted 2018-02-13 (Actual); Status verified 2005-03

CONDITIONS: Low Back Pain; Spondylolisthesis; Spinal Stenosis; Intervertebral Disc Displacement
Keywords: Spine; Lumbar spine; Spinal fusion; Low back pain; Fusion cage; Posterior lumbar interbody fusion; Bioresorbable; Peek
MeSH Terms: conditions — Low Back Pain; Spondylolisthesis; Spinal Stenosis; Intervertebral Disc Displacement

INTERVENTIONS:
Device: Lumbar Interbody Fusion

SUMMARY:
Lumbar spinal fusion is commonly performed as a "last resort" in patients with chronic low back pain caused by degenerative changes and instability of the spine. The aim of this study is to compare two fusion devices, which are used in spinal surgery in order to promote the fusion of two lumbar vertebrae.

DETAILED DESCRIPTION:
Lumbar spinal fusion is commonly performed as a "last resort" in patients with chronic low back pain caused by degenerative changes and instability of the spine. The surgical treatment involves the removal of an intervertebral disc, and subsequently the union of the two adjacent intervertebral bodies, such that a bony connection is formed within time after surgery. Lumbar spinal fusion is being performed with increasing frequency. Many interbody fusion methods have been described. In recent years, several types of fusion cages have been developed. These cages are made of various materials: titanium, stainless steel, carbon fiber or polyethylethylketone (Peek). Fusion cages have been quickly integrated into orthopedic practice.

To date, no studies have been conducted that compare the efficacy of nonresorbable and bioresorbable fusion cage devices. In this study the surgical and clinical outcomes are compared of patients with degenerative lumbar spine disorders who undergo lumbar fusion with a nonresorbable versus a bioresorbable fusion cage. Patients with lumbar spinal disorders will be recruited from several European centers and randomly allocated to one of the two intervention groups. In both treatment groups lumbar spinal fusion is performed using a standardized technique.

Patients will be evaluated during two years post-operatively. During this follow up period, the clinical outcome and fusion parameters will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Both genders, age between 18 and 70 years
* Chronic low back pain (> 3 months) with or without leg pain but no signs of motor loss
* Based on clinical history, physical examination, and radiographic signs, pain interpreted as emanating from L4-L5 or L5-S1
* Symptoms refractory to conservative treatment for at least 3 months
* Evidence of degenerative changes at L4-L5 or L5-S1 (spondylosis) on plain radiographs and/or CT scan, and/or MRI. The pathology should be predominant on one level.
* Single-level Posterior Lumbar Interbody Fusion surgery (PLIF) is indicated by the spine surgeon
* Additional posterior fixation is mandatory
* Use of autograft of the iliac crest is possible
* Ability to provide informed consent

Exclusion Criteria:

* Previous lumbar spinal fusion
* All other previous spinal surgery except for successful removal of a herniated disc more than 2 years before entering the study
* Symptomatic degenerative disc disorder at more than one lumbar level
* Pregnancy or intention to become pregnant during the two year study
* Ongoing psychiatric illness
* Evidence of alcohol and/or drug abuse
* Inability to complete the questionnaires
* Inability to walk independently
* Other indications than degenerative spinal disorders including a metabolic bone disease, osteoporosis, infection, old fracture, inflammatory process, or neoplasm
* Obvious painful and disabling arthritic hip joints

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102
Dates: Start 2004-10; Study Completion 2006-05

PRIMARY OUTCOMES:
Acquired fusion
Clinical outcome

SECONDARY OUTCOMES:
Safety and complications

CONTACTS AND LOCATIONS:
Overall Officials: P.I.J.M. Wuisman, MD, PhD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (4):
- Germany (2):
  - BG Unfallklinik Halle, Klinik für Neurochirurgie, Halle
  - Universität Rostock, Neurochirurgie, Rostock
- Netherlands (2):
  - VU University Medical Center, Amsterdam
  - Leids Universitair Medisch Centrum, Leiden

REFERENCES:
- [Background] Vaccaro AR, Singh K, Haid R, Kitchel S, Wuisman P, Taylor W, Branch C, Garfin S. The use of bioabsorbable implants in the spine. Spine J. 2003 May-Jun;3(3):227-37. doi: 10.1016/s1529-9430(02)00412-6. PMID 14589204
- [Background] Tunc DC, van Dijk M, Smit T, Higham P, Burger E, Wuisman P. Three-year follow-up of bioabsorbable PLLA cages for lumbar interbody fusion: in vitro and in vivo degradation. Adv Exp Med Biol. 2004;553:243-55. doi: 10.1007/978-0-306-48584-8_19. No abstract available. PMID 15503461
- [Background] Smit TH, Muller R, van Dijk M, Wuisman PI. Changes in bone architecture during spinal fusion: three years follow-up and the role of cage stiffness. Spine (Phila Pa 1976). 2003 Aug 15;28(16):1802-8; discussion 1809. doi: 10.1097/01.BRS.0000083285.09184.7A. PMID 12923466
- [Background] van Dijk M, Smit TH, Arnoe MF, Burger EH, Wuisman PI. The use of poly-L-lactic acid in lumbar interbody cages: design and biomechanical evaluation in vitro. Eur Spine J. 2003 Feb;12(1):34-40. doi: 10.1007/s00586-002-0458-y. Epub 2002 Sep 6. PMID 12592545
- [Background] van Dijk M, Smit TH, Burger EH, Wuisman PI. Bioabsorbable poly-L-lactic acid cages for lumbar interbody fusion: three-year follow-up radiographic, histologic, and histomorphometric analysis in goats. Spine (Phila Pa 1976). 2002 Dec 1;27(23):2706-14. doi: 10.1097/00007632-200212010-00010. PMID 12461397
- [Background] Wuisman PI, van Dijk M, Smit TH. Resorbable cages for spinal fusion: an experimental goat model. J Neurosurg. 2002 Nov;97(4 Suppl):433-9. doi: 10.3171/spi.2002.97.4.0433. PMID 12449197
- [Background] van Dijk M, Tunc DC, Smit TH, Higham P, Burger EH, Wuisman PI. In vitro and in vivo degradation of bioabsorbable PLLA spinal fusion cages. J Biomed Mater Res. 2002;63(6):752-9. doi: 10.1002/jbm.10466. PMID 12418020
- [Background] Wuisman PI, van Dijk M, Smit TH. Resorbable cages for spinal fusion: an experimental goat model. Orthopedics. 2002 Oct;25(10 Suppl):s1141-8. doi: 10.3928/0147-7447-20021002-04. PMID 12401024
- [Background] van Dijk M, Smit TH, Sugihara S, Burger EH, Wuisman PI. The effect of cage stiffness on the rate of lumbar interbody fusion: an in vivo model using poly(l-lactic Acid) and titanium cages. Spine (Phila Pa 1976). 2002 Apr 1;27(7):682-8. doi: 10.1097/00007632-200204010-00003. PMID 11923659
- [Background] Toth JM, Estes BT, Wang M, Seim HB 3rd, Scifert JL, Turner AS, Cornwall GB. Evaluation of 70/30 poly (L-lactide-co-D,L-lactide) for use as a resorbable interbody fusion cage. J Neurosurg. 2002 Nov;97(4 Suppl):423-32. doi: 10.3171/spi.2002.97.4.0423. PMID 12449196
- [Background] Toth JM, Wang M, Scifert JL, Cornwall GB, Estes BT, Seim HB 3rd, Turner AS. Evaluation of 70/30 D,L-PLa for use as a resorbable interbody fusion cage. Orthopedics. 2002 Oct;25(10 Suppl):s1131-40. doi: 10.3928/0147-7447-20021002-03. PMID 12401023
- [Background] Vaccaro AR, Robbins MM, Madigan L, Albert TJ, Smith W, Hilibrand AS. Early findings in a pilot study of anterior cervical fusion in which bioabsorbable interbody spacers were used in the treatment of cervical degenerative disease. Neurosurg Focus. 2004 Mar 15;16(3):E7. doi: 10.3171/foc.2004.16.3.8. PMID 15198495
- [Background] Lippman CR, Hajjar M, Abshire B, Martin G, Engelman RW, Cahill DW. Cervical spine fusion with bioabsorbable cages. Neurosurg Focus. 2004 Mar 15;16(3):E4. doi: 10.3171/foc.2004.16.3.5. PMID 15198492
- [Background] Krijnen MR, Smit TH, Strijkers GJ, Nicolay K, Pouwels PJ, Wuisman PI. The use of high-resolution magnetic resonance imaging for monitoring interbody fusion and bioabsorbable cages: an ex vivo pilot study. Neurosurg Focus. 2004 Mar 15;16(3):E3. doi: 10.3171/foc.2004.16.3.4. PMID 15198491
- [Background] Robbins MM, Vaccaro AR, Madigan L. The use of bioabsorbable implants in spine surgery. Neurosurg Focus. 2004 Mar 15;16(3):E1. doi: 10.3171/foc.2004.16.3.2. PMID 15198489